CLINICAL TRIAL: NCT02620904
Title: Mifepristone Induction for Fetal Demise, a Randomized Control Trial
Brief Title: Mifepristone Induction for Fetal Demise
Acronym: MIFD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to recruit. Projected completion was 2018 however, enrollment and recruitment were difficult. The study was terminated due to inability to enroll.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Atrio, principal investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-5689
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Intrauterine Fetal Demise; Fetal Death
Keywords: mifepristone; randomized controlled trial; vaginal delivery; progesterone receptor modulator; induction of labor
MeSH Terms: conditions — Stillbirth; Fetal Death | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mifepristone (Active Comparator): following informed consent women will be randomized and the mifepristone group will take 200 mg by mouth immediately prior to induction of labor for fetal demise on labor and delivery
  Interventions: Drug: Mifepristone
- placebo pill (Placebo Comparator): following informed consent women will be randomized and the placebo group will take a placebo pill by mouth (similar in properties to the mifepristone group, but it will lack any active drug) immediately prior to induction of labor for fetal demise on labor and delivery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mifepristone
  Other Names: RU486, RU46, mifeprex, mifegen
  Arms: mifepristone
Drug: placebo
  Arms: placebo pill

SUMMARY:
Methods: Double blinded, randomized controlled trial with 1:1 allocation of mifepristone or placebo at initiation of induction of labor for fetal demise 20 weeks estimated gestational age or greater.

Hypothesis: Mifepristone will expedite time to delivery of fetus among demise patients, when compared to placebo, and in conjunction with other pharmacologic methods for induction of labor.

Expected outcomes: The addition of a progesterone receptor modulator will expedite time to delivery of the fetus and ultimately improve the experience associated with induction of labor for fetal demise.

DETAILED DESCRIPTION:
The investigators propose a double blinded, randomized, placebo-controlled clinical trial at the time of initiation of induction of labor for fetal demise at 20 weeks gestational age or greater.

1. Diagnose fetal demise: confirm absence of fetal heart motion by attending physician as per the institutional standards and protocols.
2. Confirm gestational age at presentation to labor and delivery based on available medical records and/or ultrasonography as per standard practice and institutional protocols.
3. Based on inclusion and exclusion criteria potential participants will be informed about the research, offered the opportunity to contribute, and trained research staff will complete the informed consent process. After documentation of consent and discussion of the research as indicated the participants will be randomized to the intervention or control arm. Both groups will receive emotional and physical support with induction of labor as per practice guidelines and standard of care by Montefiore physicians, faculty and staff irrespective of participation or assignment.
4. Interventional Arm: Ingest 200mg tab of mifepristone orally. This will coincide with or be implemented prior to the initiation of the induction of labor plan as delineated by the attending physician. The timing will be sensitive to the needs of the participant and the labor and delivery room staff.
5. Control Arm: Ingest a placebo tab orally with similar physical properties. This will coincide with or be implemented prior to the initiation of the induction of labor plan as delineated by the attending physician. The timing will be sensitive to the needs of the participant and the labor and delivery room staff.
6. Montefiore protocol for induction of labor: will follow institutional standards.
7. Data: Patient data will be collected by the Labor and Delivery staff via electronic medical record or paper record that will be scanned into the electronic medical record. The investigators will use data abstraction tools to collect information such as time of medication administration, medications administered, time of delivery of fetus, duration of admittance to labor and delivery, and postpartum course, or complications from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Intrauterine fetal death as confirmed by absence of cardiac motion on ultrasound by Attending physician at the time of admission to the hospital.
2. Estimated gestational age greater than 20 weeks
3. Hemodynamically stable and appropriate for induction of labor as per primary clinical health team in house
4. Women with one prior low transverse cesarean delivery

Exclusion Criteria:

1. History of 2 or more low transverse cesarean deliveries
2. Prior classical cesarean delivery
3. History of abdominal myomectomy
4. Known or suspected allergic reaction to mifepristone
5. Known or suspected adrenal gland disease
6. Known or suspected bleeding diatheses or coagulopathies
7. Known or suspected use of QTc-prolonging medication
8. Known maternal medical or physical conditions that prohibits vaginal delivery

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Atrio, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone: following informed consent women will be randomized and the mifepristone group will take 200 mg by mouth immediately prior to induction of labor for fetal demise on labor and delivery
  Mifepristone
- Placebo Pill: following informed consent women will be randomized and the placebo group will take a placebo pill by mouth (similar in properties to the mifepristone group, but it will lack any active drug) immediately prior to induction of labor for fetal demise on labor and delivery
  placebo
Period: Overall Study
Arm/Group | Mifepristone | Placebo Pill
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo Pill | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery of Fetus
Description: From the initiation of medical therapy for induction to delivery of fetus, assessed up to 36 hours
Time Frame: From the initiation of medical therapy for induction to delivery of fetus, assessed up to 36 hours
Measure: Mean (Full Range); unit: hours
Arm/Group | Mifepristone | Placebo Pill
Number analyzed (Participants) | 4 | 5
hours | 14 [3 to 27] | 20 [2 to 25]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during hospitalization, an average of 3 days
Arm/Group | Mifepristone | Placebo Pill
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Due to difficulty with recruitment the study was unable to be completed in the projected time frame. Despite efforts to enhance recruitment and extending the study duration very few persons were enrolled. Due to the limited enrollment no conclusions can be ascertained about the impact of mifepristone on the induction of labor in this setting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02620904/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02620904/ICF_001.pdf